CLINICAL TRIAL: NCT06162169
Title: A Single-center, Non-randomized, Open-lable, Self-controlled Clinical Trial to Evaluate JAB-21822 Drug-drug Interactions in Healthy Subjects
Brief Title: A Clinical Trial to Evaluate JAB-21822 Drug-drug Interactions in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allist Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: JAB-21822-1010
Record Dates: First submitted 2023-11-29; First posted 2023-12-08 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-06

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Itraconazole; Omeprazole; Midazolam; Rosuvastatin Calcium; Digoxin; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- JAB-21822+Itraconazole (Experimental)
  Interventions: Drug: JAB-21822; Drug: Itraconazole
- JAB-21822+ Rifampicin (Experimental)
  Interventions: Drug: JAB-21822; Drug: Rifampicin
- JAB-21822+ Omeprazole (Experimental)
  Interventions: Drug: JAB-21822; Drug: Omeprazole
- Dazolam , Rosuvastatin calcium and digoxin with JAB-21822 (Experimental)
  Interventions: Drug: JAB-21822; Drug: Midazolam , Rosuvastatin calcium and digoxin

INTERVENTIONS:
Drug: JAB-21822 — JAB-21822 was administered orally
Drug: Itraconazole — Itraconazole was administered orally
  Arms: JAB-21822+Itraconazole
Drug: Omeprazole — Omeprazole was administered orally
  Arms: JAB-21822+ Omeprazole
Drug: Midazolam , Rosuvastatin calcium and digoxin — Midazolam , Rosuvastatin calcium and digoxin was administered orally
  Arms: Dazolam , Rosuvastatin calcium and digoxin with JAB-21822
Drug: Rifampicin — Rifampicin was administered orally
  Arms: JAB-21822+ Rifampicin

SUMMARY:
This is a phase I study to evaluate drug-drug interactions (DDIs) of JAB-21822 as a perpetrator combined with midazolam , rosuvastatin, and digoxin and to evaluate DDIs of JAB-21822 as a victim combined with itraconazole， rifampicin， and omeprazole in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ；Healthy subjects aged 18 to 50 years (including both ends) at the time of signing informed consent
2. Male subjects weighed ≥50kg, female subjects weighed ≥45kg, body mass index (BMI) was between 19.0 and 26.0kg/m2, BMI= weight (kg)/height 2 (m2), including boundary values.
3. Subjects voluntarily signed written informed consent and were able to communicate well with the investigator

Exclusion Criteria:

1. History of severe systemic diseases, history of liver and kidney insufficiency, history of mental illness, history of drug dependence;
2. Patients with a history of interstitial pneumonia, pulmonary fibrosis or other interstitial lung diseases who were not eligible for admission by the investigators;
3. Have a history of dysphagia or any gastrointestinal disease that affects drug absorption, and have digestive diseases (such as peptic ulcer, pancreatitis, colitis, etc.) within 3 months before the first dose;
4. The investigator believes that the subject has any other circumstances that make him or her unfit to participate in this clinical trial

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2023-11-25 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Observed maximum concentrations (Cmax )of JAB-21822 | approximately 10 days
Area under the concentration versus time curve from dose to the last quantifiable concentration (AUC0-t) of JAB-21822 | approximately 10 days
Area under the concentration versus time curve from dose to infinity (AUC0-∞) of JAB-21822 | approximately 10 days
Observed maximum concentrations (Cmax )of midazolam, rosuvastatin, and digoxin | approximately 10 days
Area under the concentration versus time curve from dose to the last quantifiable concentration (AUC0-t) of midazolam, rosuvastatin, and digoxin | approximately 10 days
Area under the concentration versus time curve from dose to infinity (AUC0-∞) of midazolam, rosuvastatin, and digoxin | approximately 10 days

CONTACTS AND LOCATIONS:
Overall Officials: He Qing B.Pharm, Principal Investigator — Beijing Gaobo Hospital
Locations (1):
- Beijing GoBroad Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No